CLINICAL TRIAL: NCT06219785
Title: Low-intensity Shockwave Therapy for Post-radical Prostatectomy Erectile Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Since the study opened for enrollment on June 6, 2023, we have enrolled only 5 participants, despite our goal of 100 participants over an 18-month period.
  Several factors have contributed to this decision.
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Brian Miles, Brian J Miles MD, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00037405
Record Dates: First submitted 2023-09-08; First posted 2024-01-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Intervention Model Description: Following completion of the 3-month follow-up visit, subjects will be unblinded. Subjects who received the Placebo/control treatment will be offered treatment using the active device applicator.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active (Active Comparator): 1. Patient lies down with legs extended.
  2. In order to get a proper transmission, a drop of silicone oil is applied on the anatomical stand-off before putting the ring.
  3. Connect the headpiece to the ring.
  4. Apply ultrasound gel for proper energy transmission on the shaft of the penis
  5. 1500 shocks to the lateral penile shaft (distal, mid, and proximal penile shaft), 500 impulses in each area, for a total of 1500 shocks along the penis
  6. Duration of the procedure: approximately 30 minutes
  Interventions: Device: Low-Intensity Shockwave therapy (LiSWT)
- Control (Sham Comparator): 1. Patient lies down with legs extended.
  2. In order to get a proper transmission, a drop of silicone oil is applied on the anatomical stand-off before putting the ring.
  3. Connect the headpiece to the ring.
  4. Apply ultrasound gel for proper energy transmission on the shaft of the penis
  5. 1500 shocks to the lateral penile shaft (distal, mid, and proximal penile shaft), 500 impulses in each area, for a total of 1500 shocks along the penis
  6. Duration of the procedure: approximately 30 minutes
  Interventions: Device: Low-Intensity Shockwave therapy (LiSWT)

INTERVENTIONS:
Device: Low-Intensity Shockwave therapy (LiSWT) — Participants will receive once-a-week LiSWT treatments of 0.2 mJ/ mm² over the lateral penile shaft (distal, mid, and proximal penile shaft), 500 impulses in each area, for a total of 1500 shocks along the penis once a week for six weeks, with a total of 6 treatments once a week.

SUMMARY:
This research study is trying to determine if Low-Intensity shock wave therapy (LiSWT) is safe and effective in patients with symptoms of erectile dysfunction (ED) after radical prostatectomy.

DETAILED DESCRIPTION:
Participants will be randomized to the active treatment group or the control/placebo group.

All patients on active treatment will receive Low-Intensity shock wave treatment. Participants assigned to the control group will receive the treatment using a sham applicator. The placebo group will receive the same treatment as the active group, but the transducer used for shock wave treatment will be capped, meaning that no shock waves will be transmitted to the penis.

Participants on active shock wave treatment will receive once a week Low-Intensity shock wave treatments of 0.2 mJ/ mm² over the lateral penile shaft (distal, mid, and proximal penile shaft), 500 impulses in each area, for a total of 1500 shocks along the penis once a week for six weeks, with a total of 6 treatments once a week.

ELIGIBILITY:
Inclusion Criteria:

1. Men age 45-70 who had robotic prostatectomy within 6 to 18 months
2. Documented nerve sparing during radical prostatectomy procedure
3. Mild to moderate ED after prostatectomy
4. IIEF score > 18 before surgery
5. Testosterone level > 300 mg/dl post-surgery
6. Sexually active

Exclusion Criteria:

1. Prior penile surgery
2. Lesions or active infections on the penis or perineum
3. Anatomical abnormalities in the genitalia or pelvic region
4. Unwilling to remove piercing from genital region
5. Post radical prostatectomy complications that could impact safety or effectiveness of ESWT (hematoma, unresolved anastomotic leak)
6. Previous or scheduled treatment with pelvic radiotherapy and/or androgen deprivation therapy
7. Anticoagulant medication (except acetylsalicylic acid up to 80 mg daily).
8. Any other condition that would prevent the patient from completing the study, as judged by the PI

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of LiSWT in participants with mild to moderate erectile dysfunction post-prostatectomy with the International Index of Erectile Function questionnaire. | 4 months
  The International Index of Erectile Function is a multidimensional scale that can be used to evaluate ED. It addresses the most relevant aspects of male sexual function. It involves five questions with a scale report from 0 to 5, 5 being the best value.
To assess the effectiveness of LiSWT in participants with mild to moderate erectile dysfunction post-prostatectomy with the Erectile Hardness Score questionnaire. | 4 months
  The Erection Hardness Score is a self-reported tool that measures the hardness of an erection.
  It involves a scale report from 0 to 4, 4 being the best quality of erection.

SECONDARY OUTCOMES:
To determine whether LiSWT improves the Peak systolic velocity in the Duplex Doppler Ultrasound. | 4 months
  A hemodynamic parameter commonly used in Duplex Doppler Ultrasound is Peak systolic velocity. A value of 30 cm/s or greater indicates arterial competence. The higher the parameters, the better the response to the therapy.
To determine whether LiSWT improves the Resistive index in the Duplex Doppler Ultrasound. | 4 months
  The second hemodynamic parameter commonly used in Duplex Doppler Ultrasound is the Resistive Index. A value greater than 0.90% would indicate a state of normality. The higher the parameters, the better the response to the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Miles, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist, Houston, Texas, United States